CLINICAL TRIAL: NCT05827939
Title: Association of Phenotypic Age and Antibody Titers Among SARS-Co-V2 Infected Patients and Vaccinated Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, JENG-HOW YANG, Professor Attending Physicians, Chang Gung Memorial Hospital
Other Study IDs: CMRPVVM0151
Record Dates: First submitted 2023-04-24; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Neutralizing antibody; Spike antibody; Cognitive function; long-COVID; Vaccine efficacy
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — keep plasma with five years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SARS-CoV-2 Infection: Participants from individuals with SARS-CoV-2 Infection .
  Interventions: Other: Covid19 Vaccination dose
- SARS-CoV-2 non-infection with vaccination: Participants after the second dose covid19 vaccination from individuals without SARS-CoV-2 infection.
  Interventions: Other: Covid19 Vaccination dose
- SARS-CoV-2 non-infection without vaccination: Participants get covid19 vaccination below 2 dose from individuals without SARS-CoV-2 infection.
  Interventions: Other: Covid19 Vaccination dose

INTERVENTIONS:
Other: Covid19 Vaccination dose — Participants above or below 2 dose Covid19 Vaccination

SUMMARY:
Defining the antibody response to SARS-CoV-2 will be essential for understanding disease progression, long-term immunity, and vaccine efficacy. Investigators designed a study investigating the neutralizing antibody response among post-infected and post-vaccinated individuals to determine how the spike protein neutralizing antibody correlates with natural infection and vaccination and how mutations of viral strains affect associated antibodies. New Taipei City Municipal TuCheng Hospital established a special infectious pneumonia ward in May 2021 to treat patients infected with symptomatic SARS-CoV-2 patients. During the period, 97 patients were admitted and enrolled. In light of the current timing of the pandemic, most published serological studies are predominantly cross-sectional or, at most, include a longitudinal follow-up. Cognitive function and PhenoAgeAccel will be examined for SARS-CoV-2 N and S titers decline trend analysis to correlate long-COVID brain fog or early decline of N and S antibodies.Therefore, investigators designed a three-year longitudinal study to detect patients' SARS-CoV-2 neutralizing and spike antibodies.

DETAILED DESCRIPTION:
Coronaviruses are a diverse group of viruses infecting many different animals, and th can cause mild to severe respiratory infections in humans. At the end of 2019, a novel coronavirus designated as SARS-CoV-2 emerged in Wuhan, China, and caused an outbreak of unusual viral pneumonia. Being highly transmissible, this novel coronavirus disease, also known as coronavirus disease 2019 (COVID-19), has spread fast worldwide. It has overwhelmingly surpassed SARS and MERS regarding both the number of infected people and the spatial range of epidemic areas. The ongoing outbreak of COVID-19 has posed an extraordinary threat to global public health.

Studies in large cohorts of SARS-CoV-2 infected individuals indicate that antibodies to the receptor-binding domain (RBD) of the viral spike glycoprotein appear within the first three weeks from symptoms onset, and IgG and/or IgA seroconversion occurs either sequentially or simultaneously with the appearance of IgM. Studies showed anti-RBD IgG in 95% of COVID-19 patients by the fourth week from symptom onset and observed that these antibodies increased throughout follow-up until the third-month post-hospital discharge. Moreover, the early presence of anti-RBD IgG and anti-spike IgA positively correlated with patient survival and reduced persistence of SARS-CoV-2 RNA in nasopharyngeal swabs, respectively. The spike glycoprotein mediates entry into target cells via the ACE2 receptor. Clinical trials with monoclonal antibodies (mAbs) against its RBD decreased viral load in patients with recently diagnosed mild/moderate COVID-19.

Furthermore, anti-spike neutralizing antibodies (nAbs) produced by COVID-19 patients can block viral infection of human cells in vitro and counter viral replication in vivo. However, the impact of nAbs on the COVID-19 course is still controversial, with some studies even suggesting either a detrimental role for nAbs in disease progression or finding no nAbs differences among hospitalized patients who subsequently experienced varying disease outcomes. Whether SARS-CoV-2 nAbs decline at a similar pace is yet to be conclusively established.

Defining the antibody response to SARS-CoV-2 will be essential for understanding disease progression, long-term immunity, and vaccine efficacy. Investigators designed a study investigating the neutralizing antibody response among post-infected and post-vaccinated individuals to determine how the spike protein neutralizing antibody correlates with natural infection and vaccination and how mutations of viral strains affect associated antibodies. New Taipei City Municipal TuCheng Hospital established a special infectious pneumonia ward in May 2021 to treat patients infected with symptomatic SARS-CoV-2 patients. During the period, 97 patients were admitted and enrolled. In light of the current timing of the pandemic, most published serological studies are predominantly cross-sectional or, at most, include a longitudinal follow-up. Cognitive function and PhenoAgeAccel will be examined for SARS-CoV-2 N and S titers decline trend analysis to correlate long-COVID brain fog or early decline of N and S antibodies.

Therefore, investigators designed a three-year longitudinal study to detect participantss' SARS-CoV-2 neutralizing and spike antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 20 yrs
2. Evidenced COVID-19 infeciton by PCR sequening or commercial IVD rapid test kits. (stratified by infection periods, before 2022 vs. in 2022)
3. Clealry understand the study protocol, blood drawing, organ function survey, phenoage and phenoageAccel exams and cognitive functional evaluation.
4. Agree with regular follow-up as the protocol designs

Exclusion Criteria:

1. Refuse any blood draw or follow-up schedule
2. Refuse at any time
3. The PIs judges that the patient is no longer suitable to continue the study follow-up
4. Death

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Serum samples were obtained from 3 groups of participants based on every 3-month interval. At TuCheng Hospital, infected convalescent participants were enrolled 14 days after symptom onset as the first group. Deidentified serum samples were drawn 14 days after the second dose (100-μg cohort) from participants without SARS-CoV-2 infection and post-Moderna, or AstraZeneca vaccination were enrolled as the second group. Healthy participants without SARS-CoV-2 infection were enrolled as the third group.Participants' age over 20 years old who met the enrollment criteria will be provided informed consent.These participants were prospecitvley recruited using multiple methods, including advertisements on the hospital ward, COVID-19 special clinics.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
SARS COVID N Ab trends among different subgroups | baseline
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID N Ab trends among different subgroups | 3 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID N Ab trends among different subgroups | 6 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID N Ab trends among different subgroups | 9 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID N Ab trends among different subgroups | 12 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID S Ab trends among different subgroups | baseline
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID S Ab trends among different subgroups | 3 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID S Ab trends among different subgroups | 6 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID S Ab trends among different subgroups | 9 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups
SARS COVID S Ab trends among different subgroups | 12 month
  Participants' SARS-CoV-2 neutralizing antibody measure among different subgroups

SECONDARY OUTCOMES:
SARS COVID N Ab trends among different baseline PhenoAge scores | baseline
  Hematology measure associated with PhenoAge scores
SARS COVID N Ab trends among different baseline PhenoAge scores | 3 month
  Hematology measure associated with PhenoAge scores
SARS COVID N Ab trends among different baseline PhenoAge scores | 6 month
  Hematology measure associated with PhenoAge scores
SARS COVID N Ab trends among different baseline PhenoAge scores | 9 month
  Hematology measure associated with PhenoAge scores
SARS COVID N Ab trends among different baseline PhenoAge scores | 12 month
  Hematology measure associated with PhenoAge scores
SARS COVID S Ab trends among different baseline PhenoAge scores | baseline
  PhenoAge scores relation physiology measure
SARS COVID S Ab trends among different baseline PhenoAge scores | 3 month
  Hematology measure associated with PhenoAge scores
SARS COVID S Ab trends among different baseline PhenoAge scores | 6 month
  Hematology measure associated with PhenoAge scores
SARS COVID S Ab trends among different baseline PhenoAge scores | 9 month
  Hematology measure associated with PhenoAge scores
SARS COVID S Ab trends among different baseline PhenoAge scores | 12 month
  Hematology measure associated with PhenoAge scores

CONTACTS AND LOCATIONS:
Overall Officials: Jeng-How Yang, Study Director — Division of Infections Disease, Chang Gung Memorial Hospital
Locations (1):
- TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided